CLINICAL TRIAL: NCT02446678
Title: The Use Of PillCam Esophagus In Triaging Patients Presented With Upper Gastrointestinal Bleeding
Brief Title: Use of PillCam ESO2 in Triaging Patients Present With Upper GIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ESO2
Record Dates: First submitted 2015-05-12; First posted 2015-05-18 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Gastrointestinal bleeding; emergency department; PillCam ESO2
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsule group: PillCam ESO2 (Active Comparator): Perform capsule endoscopy and esophagogastroduodenoscopy will be preformed within 24 hours after capsule ingestion
  Interventions: Device: PillCam ESO2
- Standard group (No Intervention): Perform standard esophagogastroduodenoscopy

INTERVENTIONS:
Device: PillCam ESO2 — Capsule endoscopy
  Arms: Capsule group: PillCam ESO2

SUMMARY:
Background

* Patients presented to hospital with coffee ground vomiting and black stool may not be actually having upper gastrointestinal bleeding (UGIB)
* Hospital admission can be avoided if serious UGIB can be excluded
* To date, the only useful tool to triage patient for hospital admission in UGIB is by using clinical score such as Rockall score or Blatchford score
* These scores are cumbersome and only exclude the most benign cases, but they are not useful in differentiating those who needs intervention
* In our pilot study, investigators found that capsule endoscopy can be used to identify patients with fresh blood and real coffee ground substance in the stomach and it is superior to nasogastric tube
* Most of UGI lesions leading to bleeding can be diagnosed by capsule endoscopy

Objectives The current study is designed

1. to validate capsule endoscopy is an effective method in identifying patients with UGIB
2. to study whether the capsule endoscopy can reduce requirement of hospital admission in patients with suspected UGIB
3. to study if capsule endoscopy can help to identify patients with UGIB that may require urgent (within 24 hours) endoscopy and intervention
4. to study the cost-effectiveness of capsule endoscopy being used as a triaging tool in the management of UGIB
5. to compare the effectiveness of capsule endoscopy against Blatchford score in identifying patients with UGIB that may require endoscopic intervention.

DETAILED DESCRIPTION:
Hypothesis PillCam Esophagus is effective in identifying genuine UGIB and hence able to reduce hospital admission due to unsubstantiated UGIB cases

Methodology

* Patients presented to the Accident & Emergency Department (A&ED) of the Prince of Wales Hospital Hong Kong with symptoms suggestive of UGIB will be recruited into this study
* Patients will receive the following tests

  * Complete blood count
  * Coagulation profile
  * Renal and liver function tests
  * Hourly BP, Pulse up to 6 hours
  * Glasgow Blatchford score calculated on admission
* Randomization

  * Capsule Group: Capsule Endoscopy (CE) by using PillCam Esophagus (PillCam ESO) OR
  * Standard group: Hospitalization and Standard of Care
* The video in capsule endoscopy will be read by trained personnel who have undergone at least one hour lecture about realtime reviewing.
* Legally a patient has to be signed off by a clinician within 6 hours. The finding of fresh blood or coffee ground will be documented. Upper GI pathology that may lead to bleeding will also be recorded.

Capsule Endoscopy (CE) After confirming patient has been fasted for at least 5 hours, the subject ingested the PillCam® ESO 2 (Given Imaging Ltd., Yoqneam, Israel) (PillCam ESO) using the Simplified Ingestion Procedure.

Thirty to sixty minutes prior to capsule ingestion, each subject received a single dose of intravenous Maxolon 10mg. Intravenous Maxolon, through its motilin receptor agonist effect, has been shown to promote gastric motility and improve visualization of the gastric mucosa at endoscopy. Moreover, use of Maxolon was thought to facilitate the capsule entering the duodenum.

Using the REAL time viewer, UGI tract images (esophagus to the second portion of the duodenum) were obtained in real time at the patient's bedside. The video images that are transmitted by the PillCam ESO 2 are displayed in real time on the tablet computer screen.

Each subject is also fitted with and wore the standard CE sensor array and data recorder so that a full-length CE video recording can be obtained for subsequent capsule workstation downloading and complete review.

Other demographic data and parameters for Blatchford score calculation will be collected. 10 ml of blood will be taken for routine blood checking. Patients will receive standard care according to EGD findings.

ELIGIBILITY:
Inclusion Criteria:

Individual aged ≥ 18 years presenting to the emergency department with acute, overt UGIB defined as coffee ground vomiting and/or melena

Exclusion Criteria:

* UGIB with hemodynamic shock (BP<90mmHg and pulse>120 per minutes) requiring urgent endoscopy,
* UGIB with fresh hematemesis requiring urgent endoscopy
* dysphagia, odynophagia, swallowing disorder, Zencker's diverticulum, suspected bowel obstruction or bowel perforation,
* prior bowel obstruction, gastroparesis or known gastric outlet obstruction, Crohn's disease, past GI tract surgery.
* presence of an electromedical device (pacemaker or internal cardiac defibrillator),
* altered mental status (e.g., hepatic encephalopathy) that would limit patient ability in swallowing the capsule, pregnancy and/or lactating, allergy to conscious sedation medications, allergy to Maxolon, unwillingness to swallow the capsule, patient expected to undergo Magnetic Resonance Imaging examination within 7 days of ingesting the capsule, patient on medications that may coat the upper GI tract such as antacids or sucralfate, or inability to provide written informed consent.
* Allergy to Maxolon
* Patients with known Esophageal Varices or Gastric Varices with or without prior bleeding episodes
* Known upper/ lower GI cancer (eg, cancer of esophagus, stomach, small bowel, colon) or hepatocellular carcinoma or pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The number of patients requiring hospital admission | 24 hours
  Patients with evidence of significant bleeding will be admitted to ward and receive early endoscopy (EGD)

SECONDARY OUTCOMES:
Clinical rebleeding | 30 days
  Recurrent GI bleeding
Mortality | 30 days
  Death rate
Cost of management in different strategies | One year
  Cost of management in different strategies
Comparing the effectiveness of CE against Glasgow Blatchford score in identifying patients with UGIB that may require endoscopic intervention | 30 days
  Using Glasgow Blatchford score

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Y.L. Ching, MPH, Study Director — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung JJ, Tang RS, Ching JY, Rainer TH, Lau JY. Use of capsule endoscopy in the emergency department as a triage of patients with GI bleeding. Gastrointest Endosc. 2016 Dec;84(6):907-913. doi: 10.1016/j.gie.2016.04.043. Epub 2016 May 6. PMID 27156655